CLINICAL TRIAL: NCT02749305
Title: Comparative Effectiveness of Metabolic and Bariatric Surgical Procedures Using Patient Reported Outcome Measures (PROMs)
Brief Title: Comparative Effectiveness of Metabolic and Bariatric Surgery With PROMs
Acronym: MBSAQIP-PROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthew Hutter, Medical Director of the Codman Center, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016P000346; CER-1503-29209 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2016-03-25; First posted 2016-04-22 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Bariatric Surgery; Metabolic Surgery; Weight Reduction
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preop Metabolic & Bariatric Patients (Other): Attempted collection of patient-reported outcome measures preoperatively and annually postoperatively will occur with all metabolic and bariatric surgery patients scheduled for surgery at a participating center.
  Interventions: Other: Collection of patient-reported outcome measures
- Postop Metabolic & Bariatric Patients (Other): Attempted collection of patient-reported outcome measures annually postoperatively will occur with all metabolic and bariatric surgery patients who had surgery at a participating center within the preceding 12 months.
  Interventions: Other: Collection of patient-reported outcome measures

INTERVENTIONS:
Other: Collection of patient-reported outcome measures — Preoperative and postoperative metabolic and bariatric surgery patients will be asked to electronically complete a set of PROMs up to 21 days before surgery and annually on their surgical anniversary they will be asked to complete a postoperative PROM.

SUMMARY:
This long-term, nationwide observational data collection repository will obtain patient-reported outcomes from metabolic and bariatric surgery patients. The data will be used in conjunction with clinical outcomes to determine quality, safety, and comparative effectiveness of various metabolic and bariatric procedures.

ELIGIBILITY:
Inclusion Criteria All preoperative metabolic and bariatric surgery patients with a scheduled metabolic and bariatric surgery at a participating center are eligible for inclusion.

Postoperative metabolic and bariatric surgery patients must have had their surgery within the preceding year at a participating center.

Exclusion Criteria Metabolic and bariatric surgery patients without an already scheduled surgery date at a participating center.

Postoperative metabolic and bariatric surgery patients who are more than 1 year postop from a participating center.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11146 (Actual)
Dates: Start 2016-03; Primary Completion 2024-02 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Patient-reported PROMIS (Patient-Reported Outcomes Measurement Information System) 10 | preoperatively and annually postoperatively
  patients will be asked to complete the PROMIS (Patient-Reported Outcomes Measurement Information System) 10 survey
Patient-reported Obesity-related Problems | preoperatively and annually postoperatively
  patients will be asked to complete the Obesity-related Problems Scale
Patient-reported Obesity and Weight-loss Quality of Life | preoperatively and annually postoperatively
  patients will be asked to complete the Obesity and Weight-loss Quality of Life instrument
Patient-reported comorbidities | annually postoperatively
  patients will be asked to report their obesity-related comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greene ME, Grieco A, Evans-Labok K, Ko CY, Hutter MM. First report of outcomes from the patient-reported outcome measures program in the Metabolic and Bariatric Surgery Accreditation Quality Improvement Program. Surg Obes Relat Dis. 2024 Feb;20(2):173-183. doi: 10.1016/j.soard.2023.09.010. Epub 2023 Sep 15. PMID 37949691
- [Background] Greene ME, Goldman RE, Hutter MM. Selection of patient-reported outcomes measures for implementation in the Metabolic and Bariatric Surgery Accreditation Quality Improvement Program. Surg Obes Relat Dis. 2023 Aug;19(8):897-906. doi: 10.1016/j.soard.2023.01.031. Epub 2023 Feb 9. PMID 37037688
- [Background] Grieco A, Greene ME, Ko CY, Cohen ME, Evans-Labok K, Fraker T, Hutter MM. Evaluating agreement between clinic- and patient-reported outcomes for weight and co-morbidities at 1 year after bariatric surgery. Surg Obes Relat Dis. 2023 Apr;19(4):309-317. doi: 10.1016/j.soard.2022.10.001. Epub 2022 Oct 11. PMID 36400692